CLINICAL TRIAL: NCT04028479
Title: The Registry of Oncology Outcomes Associated with Testing and Treatment (ROOT)
Brief Title: The Registry of Oncology Outcomes Associated with Testing and Treatment
Acronym: ROOT
Status: Completed | Type: Observational
Sponsor: Taproot Health (Industry)
Responsible Party: Sponsor
Other Study IDs: ROOT
Record Dates: First submitted 2019-07-17; First posted 2019-07-22 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Adenocarcinoma; Adenocystic Carcinoma; Anal Cancer; Appendix Cancer; Brain Tumor; Glioblastoma; Astrocytoma; Bile Duct Cancer; Cholangiocarcinoma; Bladder Cancer; Bone Cancer; Synovial Sarcoma; Chondrosarcoma; Liposarcoma; Sarcoma, Kaposi; Sarcoma,Soft Tissue; Sarcoma; Osteosarcoma; CNS Cancer; Brain Stem Neoplasms; Breast Cancer; Cervical Cancer; Colorectal Cancer; Rectal Cancer; Colon Cancer; Esophageal Cancer; Esophagus Cancer; Cancer of Colon; Pancreatic Cancer; Cancer of Pancreas; Testis Cancer; Testicular Cancer; Ureter Cancer; Renal Cell Carcinoma; Kidney Cancer; Gestational Trophoblastic Tumor; Head and Neck Neoplasms; Parotid Tumor; Larynx Cancer; Tongue Cancer; Pharynx Cancer; Salivary Gland Cancer; Acute Myeloid Leukemia; Chronic Myeloid Leukemia; Acute Lymphoblastic Leukemia; Multiple Myeloma; Non Hodgkin Lymphoma; Carcinoid Tumor; Lung Cancer; Neuroendocrine Tumors; Mesothelioma; Thyroid Cancer; Parathyroid Neoplasms; Adrenal Cancer; Small Bowel Cancer; Stomach Cancer; Liver Cancer; Hepatic Cancer; Melanoma; Skin Cancer; Unknown Primary Tumors; Uterine Cancer; Fallopian Tube Cancer; Ovarian Cancer; Prostate Cancer; Vaginal Cancer; Penile Cancer; Vulvar Cancer; Waldenstrom Macroglobulinemia; Cancer, Advanced; Thymus Cancer; Nasopharyngeal Carcinoma; Multiple Endocrine Neoplasia; Pheochromocytoma; Small Cell Carcinoma; Pulmonary Carcinoma
Keywords: Precision Medicine; Molecular Sequence Data; Databases, Genetic; High-Throughput Nucleotide Sequencing; Massively-Parallel Sequencing; Observational Study; Treatment; Patient Outcome Assessment; Adaptive clinical trial; Molecular Typing; Response Rate; Progression Free Survival; Overall Survival
MeSH Terms: conditions — Adenocarcinoma; Carcinoma, Adenoid Cystic; Anus Neoplasms; Appendiceal Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Bile Duct Neoplasms; Cholangiocarcinoma; Urinary Bladder Neoplasms; Bone Neoplasms; Sarcoma, Synovial; Chondrosarcoma; Liposarcoma; Sarcoma, Kaposi; Sarcoma; Osteosarcoma; Central Nervous System Neoplasms; Brain Stem Neoplasms; Breast Neoplasms; Uterine Cervical Neoplasms; Colorectal Neoplasms; Rectal Neoplasms; Colonic Neoplasms; Esophageal Neoplasms; Pancreatic Neoplasms; Testicular Neoplasms; Ureteral Neoplasms; Carcinoma, Renal Cell; Kidney Neoplasms; Gestational Trophoblastic Disease; Head and Neck Neoplasms; Parotid Neoplasms; Laryngeal Neoplasms; Tongue Neoplasms; Pharyngeal Neoplasms; Salivary Gland Neoplasms; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Multiple Myeloma; Lymphoma, Non-Hodgkin; Carcinoid Tumor; Lung Neoplasms; Neuroendocrine Tumors; Mesothelioma; Thyroid Neoplasms; Parathyroid Neoplasms; Adrenal Gland Neoplasms; Stomach Neoplasms; Liver Neoplasms; Melanoma; Skin Neoplasms; Neoplasms, Unknown Primary; Uterine Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Vaginal Neoplasms; Penile Neoplasms; Vulvar Neoplasms; Waldenstrom Macroglobulinemia; Neoplasms; Thymus Neoplasms; Nasopharyngeal Carcinoma; Multiple Endocrine Neoplasia; Pheochromocytoma; Carcinoma, Small Cell | interventions — Molecular Diagnostic Techniques; Biological Therapy; Immunotherapy; Drug Therapy; Patient Reported Outcome Measures; Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Protocol does not require submission of samples, but catalogs location of specimens that can be requisitioned later
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Validation Cohort: Patients enrolled into the study to allow validation of a specific element, process, or endpoint. Validation will be done showing concordance with traditional interventional trial standards.
  Interventions: Diagnostic Test: Biomarker Testing (L); Drug: Systemic Treatment (T)
- Analysis Cohorts: Patient who are enrolled into the study to allow analysis to determine any association, effect, or benefit. Cohorts can be determined prospectively and/or retrospectively for data already collected, Cohorts are identified to highlight collection of information on patients who are already receiving any treatment or testing as determined by the physician and patient independent of this study. Because many analysis cohorts will be determined in patients already enrolled in the study, this group is inclusive of many different sub-groupings or specific analysis cohorts of patients.
  Interventions: Diagnostic Test: Biomarker Testing (L); Drug: Systemic Treatment (T); Other: Patient Reported Outcomes (P)
- Retrospective Chart Review Cohorts: This arm will use retrospective data obtained through systematic chart review on previously seen patients to compare, contrast, or enhance the efforts of the prospective arms. Because most RWD has been traditionally obtained through retrospective methods, this is also considered the "control arm." Data in this arm will be collected without any patient identifiers. This arm is optional.

INTERVENTIONS:
Diagnostic Test: Biomarker Testing (L) — Patients who have received biomarker testing that could affect prognosis or treatment decisions. This generally excludes testing done to assist in the diagnosis of disease or histology where there is no treatment implication from this testing.
  Other Names: Biomarker Testing; Molecular Testing; Next-generation sequencing (NGS); Multiplex molecular testing
  Groups: Analysis Cohorts; Validation Cohort
Drug: Systemic Treatment (T) — Patients who have received any treatment as part of their care. This refers to systemic treatment, but also allows other non-drug related interventions such as surgery or radiotherapy as part of the longitudinal care of the patient.
  Other Names: Biologic therapy; Targeted therapy; Immunotherapy; Chemotherapy
  Groups: Analysis Cohorts; Validation Cohort
Other: Patient Reported Outcomes (P) — Patients who have provided information about their disease, treatment course, or experience directly to the study using a patient facing tool or device.
  Other Names: Patient experience; Quality of life; Self-reporting
  Groups: Analysis Cohorts

SUMMARY:
This study is to collect and validate regulatory-grade real-world data (RWD) in oncology using the novel, Master Observational Trial construct. This data can be then used in real-world evidence (RWE) generation. It will also create reusable infrastructure to allow creation or affiliation with many additional RWD/RWE efforts both prospective and retrospective in nature.

DETAILED DESCRIPTION:
This is a master observational trial (MOT). Anyone who has been diagnosed with advanced cancer is eligible as long as they are a candidate for treatment. Each patient will receive testing and treatment as determined by patient in consultation with physician. ROOT will proceed in two directions: (1) Validation Cohorts. These patients will demonstrate the ability of the MOT to prospectively collect data using the same protocol and related documents, standardized data elements and processes, and accepted scientific endpoints; and (2) Analysis Cohorts. The modular nature of the study allows collection of RWD ranging from diagnosis only to the full treatment course of the of the patient. Patients are grouped to allow focused data collection or a specific analysis. Analysis cohorts can be created from patients already enrolled in ROOT or be defined prospectively. Because of the ongoing advancements of molecular based oncology, this trial allows a detailed focus on molecular testing as part of any cohort.

Data is reported by the group that is most qualified to provide this information and is proved, at point of care, using standardized data elements and processes. Physicians will report diagnosis, molecular characteristics, staging, disease burden, significant comorbidities, treatment response, and medical decision making. Molecular testing (reports and details) will be requested from testing laboratories. Any diagnostic films will be received digitally from the location the study was performed. Research staff assist in data entry and providing physicians needed data as part of the regular workflow to allow point-of-care reporting.

The Validation Cohorts and Analysis Cohorts may run sequentially or in parallel with each other.

ELIGIBILITY:
Inclusion Criteria:

* Patient or representative provides written informed consent
* Patient is diagnosed with advanced malignancy
* Patient is willing to be treated for this malignancy according to a plan determine by them and their physician
* patient will be willing to have regular follow up visits as part of their standard of care

Exclusion Criteria:

* patient is not a candidate or does not desire any treatment for their disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with advanced cancer is eligible for inclusion in this study. Sponsor may identity specific subsets of patients that have a specific characteristic, received a certain type of testing or treatment, or are followed for a certain time period as part of their standard of care independent of this study. These identified areas will never exclude any gender, race, or socioeconomic status.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Best overall response (BOR) - 1st line of therapy | 1st line of therapy, on average less than 1 year
  The best overall response for 1st line of therapy as determined by physician assessment
Best overall response (BOR) - 2nd line of therapy | 2nd line of therapy, on average less than 1 year
  The best overall response for 2nd line of therapy as determined by physician assessment
Best overall response (BOR) - 3rd line of therapy | 3rd line of therapy, on average less than 1 year
  The best overall response for 3rd line of therapy as determined by physician assessment
Best overall response (BOR) - 4th line of therapy | 4th line of therapy, on average less than 1 year
  The best overall response for 4th line of therapy as determined by physician assessment
Best overall response (BOR) - 5th line of therapy | 5th line of therapy, on average less than 1 year
  The best overall response for 5th line of therapy as determined by physician assessment
Progression-free survival (PFS) - 1st line of therapy | 1st line of therapy, on average less than 1 year
  The progression free survival for 1st line of therapy as determined by physician assessment
Progression-free survival (PFS) - 2nd line of therapy | 2nd line of therapy, on average less than 1 year
  The progression free survival for 2nd line of therapy as determined by physician assessment
Progression-free survival (PFS) - 3rd line of therapy | 3rd line of therapy, on average less than 1 year
  The progression free survival for 3rd line of therapy as determined by physician assessment
Progression-free survival (PFS) - 4th line of therapy | 4th line of therapy, on average less than 1 year
  The progression free survival for 4th line of therapy as determined by physician assessment
Progression-free survival (PFS) - 5th line of therapy | 5th line of therapy, on average less than 1 year
  The progression free survival for 5th line of therapy as determined by physician assessment

SECONDARY OUTCOMES:
Overall survival (OS) | through study completion, on average less than 3 years
  The overall survival of a patient from the time of being diagnosed with advanced disease until death

CONTACTS AND LOCATIONS:
Overall Officials: Razelle Kurzrock, MD, Study Chair — Moores Cancer Center at University of California at San Diego; Vivek Subbiah, MD, Principal Investigator — M.D. Anderson Cancer Center; Jennifer Johnson, MD, PhD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University; Raymond Bergan, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - Teton Cancer Institute, Idaho Falls, Idaho
  - Oncology and Hematology of South Texas, Laredo, Texas

IPD SHARING:
Plan to Share IPD: Undecided
IPD will likely be shared, but will be determined by participating clinical sites.

REFERENCES:
- [Background] Woodcock J, LaVange LM. Master Protocols to Study Multiple Therapies, Multiple Diseases, or Both. N Engl J Med. 2017 Jul 6;377(1):62-70. doi: 10.1056/NEJMra1510062. No abstract available. PMID 28679092
- [Background] Boland JF, Chung CC, Roberson D, Mitchell J, Zhang X, Im KM, He J, Chanock SJ, Yeager M, Dean M. The new sequencer on the block: comparison of Life Technology's Proton sequencer to an Illumina HiSeq for whole-exome sequencing. Hum Genet. 2013 Oct;132(10):1153-63. doi: 10.1007/s00439-013-1321-4. Epub 2013 Jun 12. PMID 23757002
- [Background] Morash M, Mitchell H, Beltran H, Elemento O, Pathak J. The Role of Next-Generation Sequencing in Precision Medicine: A Review of Outcomes in Oncology. J Pers Med. 2018 Sep 17;8(3):30. doi: 10.3390/jpm8030030. PMID 30227640
- [Background] Korphaisarn K, Kopetz S. BRAF-Directed Therapy in Metastatic Colorectal Cancer. Cancer J. 2016 May-Jun;22(3):175-8. doi: 10.1097/PPO.0000000000000189. PMID 27341594
- [Background] Sherman RE, Anderson SA, Dal Pan GJ, Gray GW, Gross T, Hunter NL, LaVange L, Marinac-Dabic D, Marks PW, Robb MA, Shuren J, Temple R, Woodcock J, Yue LQ, Califf RM. Real-World Evidence - What Is It and What Can It Tell Us? N Engl J Med. 2016 Dec 8;375(23):2293-2297. doi: 10.1056/NEJMsb1609216. No abstract available. PMID 27959688
- [Background] Kaplan RM, Chambers DA, Glasgow RE. Big data and large sample size: a cautionary note on the potential for bias. Clin Transl Sci. 2014 Aug;7(4):342-6. doi: 10.1111/cts.12178. Epub 2014 Jul 15. PMID 25043853
- [Background] AACR Project GENIE Consortium. AACR Project GENIE: Powering Precision Medicine through an International Consortium. Cancer Discov. 2017 Aug;7(8):818-831. doi: 10.1158/2159-8290.CD-17-0151. Epub 2017 Jun 1. PMID 28572459
- [Background] Dickson DJ, Pfeifer JD. Real-world data in the molecular era-finding the reality in the real world. Clin Pharmacol Ther. 2016 Feb;99(2):186-97. doi: 10.1002/cpt.300. Epub 2016 Jan 12. PMID 26565654
- [Background] Conley RB, Dickson D, Zenklusen JC, Al Naber J, Messner DA, Atasoy A, Chaihorsky L, Collyar D, Compton C, Ferguson M, Khozin S, Klein RD, Kotte S, Kurzrock R, Lin CJ, Liu F, Marino I, McDonough R, McNeal A, Miller V, Schilsky RL, Wang LI. Core Clinical Data Elements for Cancer Genomic Repositories: A Multi-stakeholder Consensus. Cell. 2017 Nov 16;171(5):982-986. doi: 10.1016/j.cell.2017.10.032. PMID 29149611